CLINICAL TRIAL: NCT00820495
Title: Effectiveness of a Web-Assisted Quitline for Smokeless Tobacco Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01CA084225 (NIH); R01CA084225 (NIH)
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Tobacco Use Disorder
Keywords: Smokeless tobacco; Chewing Tobacco; Internet; Adolescent
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Web + Phone (Experimental): Highly interactive tailored Web-based smokeless tobacco cessation program plus phone counseling
  Interventions: Behavioral: Web + Phone
- Web Only (Experimental): Highly interactive tailored Web-based smokeless tobacco cessation program
  Interventions: Behavioral: Web Only
- Phone Only (Experimental): Phone counseling intervention for smokeless tobacco cessation
  Interventions: Behavioral: Phone Only
- Control (Experimental): Usual care (initial call plus self-help materials)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Web + Phone — Web + Phone
  Other Names: web-assisted intervention; quitline; helpline
  Arms: Web + Phone
Behavioral: Web Only — Web Only
  Other Names: web-assisted intervention
  Arms: Web Only
Behavioral: Phone Only — Phone Only
  Other Names: helpline; quitline
  Arms: Phone Only
Behavioral: Usual Care — Usual Care
  Other Names: helpline; quitline
  Arms: Control

SUMMARY:
The purpose of this record is to test whether (a) participants who receive a Web-based smokeless tobacco cessation intervention will be more likely to be abstinent than participants who do not receive this intervention, and (b) whether participants who receive a telephone quitline intervention will be more likely to be abstinent than participants who are not in a quitline intervention.

DETAILED DESCRIPTION:
Many Americans engage in the habitual use of smokeless tobacco (ST), and many wish to quit but lack resources. There is a need for innovative, validated, and easily delivered low-cost interventions to facilitate ST cessation in this under-served population of tobacco users. In our current ChewFree study, we have developed a user-friendly, interactive Web-based intervention, and in a randomized trial we have shown this website to be more efficacious than a rigorous control condition that offered Web-based basic textual information on ST cessation. We now seek to extend this proven approach by marrying it with a quitline telephone counseling service that has been used with noteworthy success for smoking abstinence but has not yet been evaluated with ST users. Our 2 x 2 design and large sample size allow us to test both main effects - Web program, phone counseling - as well as explore planned comparisons to examine the value-added contribution of the Web-based intervention to phone counseling, and vice-versa.

This project takes advantage of the opportunity to conduct a study of two tobacco cessation interventions that are growing in use. The use of tobacco help lines is now almost ubiquitous, with more than 30 state and national services now being offered. The use of the Internet for health information and behavior change (including tobacco cessation) has been growing in popularity as well. The proposed project would be an extension of both lines of research, evaluating the relative efficacy of our Internet-based program, telephone counseling, and the combination of both.

We will use a multifaceted promotional plan to recruit more than 2,000 ST users. The recruitment plan builds on the collaborative marketing efforts of a state tobacco control organization and organized promotion through media mailings, on-line advertising, and direct mailing. Follow-up assessment data will be collected electronically via the Internet supplemented by telephone follow-up. Additional data will be derived from phone counselor notes and measures of website usage.

ELIGIBILITY:
Inclusion Criteria:

* current users of smokeless tobacco products (snuff or chewing tobacco)
* use of smokeless tobacco products for at least 1 year
* use of at least one tin or pouch per week
* interest in quitting all tobacco
* U.S. resident 18 years of age or older
* ability to read English
* willingness to share a phone number, e-mail, and mailing address
* use of personal Internet e-mail account at least once per week
* informed consent

Exclusion criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1683 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prolonged abstinence from all tobacco | 3 months and 6 months

SECONDARY OUTCOMES:
7-day point prevalence for smokeless tobacco use | 3 months and 6 months
7-day point prevalence for all tobacco use | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert H. Severson, PhD, Principal Investigator — Oregon Research Institute
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - Oregon Research Institute, Eugene, Oregon

REFERENCES:
- [Derived] Danaher BG, Severson HH, Zhu SH, Andrews JA, Cummins SE, Lichtenstein E, Tedeschi GJ, Hudkins C, Widdop C, Crowley R, Seeley JR. Randomized Controlled Trial of the Combined Effects of Web and Quitline Interventions for Smokeless Tobacco Cessation. Internet Interv. 2015 May 1;2(2):143-151. doi: 10.1016/j.invent.2015.02.005. PMID 25914872